CLINICAL TRIAL: NCT04587128
Title: Phase II Trial of Early-Line Anti-EGFR Therapy to Facilitate Retreatment for Select Patients With Metastatic Colorectal Cancer
Brief Title: Early-Line Anti-EGFR Therapy to Facilitate Retreatment for Select Patients With mCRC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0714; 2020-0714 (Registry Identifier: Health Science IRB); NCI-2020-06543 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); Protocol Version 6/17/2025 (Other: UW Madison)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Cetuximab; Irinotecan; IFL protocol; Bevacizumab

STUDY DESIGN:
Intervention Model Description: The study is an open label phase 2 clinical trial with 3 independent study arms conducted through the University of Wisconsin Carbone Cancer Center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: No Previous EGFR (Experimental): Participant who have not be previously exposed to anti-EGFR therapies and are in the first or second-line metastatic treatment setting.
  Panitumumab (6mg/kg) or Cetuximab 500mg (per treating physician) on day 1 and 15 of a 28-day cycle
  Interventions: Drug: Panitumumab; Drug: Cetuximab
- Cohort B: Retreatment (Experimental): Participants with treatment refractory disease who have previously benefitted (greater than or equal to 4 months ago) from anti-EGFR therapy.
  Panitumumab (6mg/kg) or Cetuximab 500mg (per treating physician) on day 1 and 15 of a 28-day cycle, +/- Irinotecan (180mg/m^2) every 2 two weeks per standard of care
  Interventions: Drug: Panitumumab; Drug: Cetuximab; Drug: Irinotecan
- Cohort C: Rechallenge (Experimental): Participants with prior FOLFOX and either no prior EGFR inhibitor or treated on Cohort A.
  Alternating Panitumumab (6mg/kg) or Cetuximab 500mg (per treating physician) and 4 cycles of FOLFIRI +/- bevacizumab
  Interventions: Drug: Panitumumab; Drug: Cetuximab; Drug: FOLFIRI Protocol; Drug: Bevacizumab

INTERVENTIONS:
Drug: Panitumumab — Epidermal growth factor receptor inhibitor, anti-neoplastic
Drug: Cetuximab — Epidermal growth factor receptor inhibitor, anti-neoplastic
Drug: Irinotecan — anti-neoplastic, chemotherapy drug
  Arms: Cohort B: Retreatment
Drug: FOLFIRI Protocol — folinic acid (also called leucovorin, calcium folinate or FA) fluorouracil (also called 5FU) irinotecan given per institutional standard (intravenously day 1 and day 15 of 28 day cycle) alternating and not concomitant with panitumumab or cetuximab
  Arms: Cohort C: Rechallenge
Drug: Bevacizumab — Bevacizumab (or biosimilar) may be administered with FOLFIRI per treating MD discretion and will be given per institutional standard (5 mg/kg intravenously day 1 and day 15 of 28 day cycle)
  Arms: Cohort C: Rechallenge

SUMMARY:
The study will use previously established doses of panitumumab or cetuximab in the metastatic setting for the treatment of unresectable colorectal cancer (CRC). It is designed to investigate an alternative treatment strategy to maximize the benefit to inhibition of epidermal growth factor receptor (EGFR) for a highly selected patient population. It will enroll 71 participants with left-sided, unresectable metastatic CRC. Participants will be on study up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information
* As determined by the enrolling physician or protocol designee, ability of the participant to understand and comply with study procedures for the entire length of the study
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
* Have a diagnosis of histologically confirmed metastatic colorectal cancer with primary tumor located beyond the splenic flexure. Histologic confirmation of a colorectal primary tumor is acceptable if accompanied by radiographic evidence of metastatic disease.

  * For Cohort A: Participants must enroll for study treatment in the first or second-line metastatic setting. Participants may receive 1 month of standard chemotherapy in the metastatic setting and still be eligible to initiate protocol therapy in the first-line setting. Adjuvant or neoadjuvant therapy does not count as a line of therapy even if given in the setting of metastatic disease (oligometastatic), unless disease recurrence was noted within 6 months of completing the last dose of the adjuvant or neoadjuvant therapy.
  * For Cohort B: Participants must have had at least stable disease (per treating physician) on a prior EGFR inhibitor containing regimen and it must be at least 4 months since the prior anti-EGFR inhibitor treatment was completed. Participants previously enrolled in Cohort A can later enroll in Cohort B should the eligibility criteria be met.
  * For Cohort C: Subjects with no prior use of irinotecan or anti-EGFRi. If patients were treated on cohort A (of this study) they can cross-over to cohort C if other eligibility criteria are met at the time of cross-over.
* Evaluable disease according to RECIST v1.1. Participants do not have to have measureable disease.
* Participants with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic.
* Demonstrate adequate organ function; all screening labs to be obtained within 7 days prior to registration. Note minimum platelet requirement differs between Cohort A and B.

  * Absolute Neutrophil Count (ANC) ≥ 1,000 / mcL
  * Platelets ≥ 50,000 / mcL (Cohort A); ≥ 50,000 mcL (Cohort B receiving only EGFRi); ≥75,000 / mcL (cohort B receiving irinotecan and EGFRi; and cohort C)
  * Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 2.0 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels > 2.0 X institutional ULN
  * Bilirubin ≤ 1.5 × ULN OR direct bilirubin ≤ ULN for subjects with bilirubin levels >1.5 x ULN
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 5 × ULN
  * Albumin ≥ 2.5 mg/dL
* Females of childbearing potential must have a negative serum pregnancy test within 7 days of registration and not be breastfeeding. Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* Tumor must be mismatch repair (MMR) proficient as determined by microsatellite instability or immunohistochemistry for MMR proteins

  * Microsatellite instability (MSI) testing must be MSI-stable or MSI-low.
  * Or IHC for MMR proteins must demonstrate intact MMR proteins.
* Baseline (prior to any anti-EGFR treatment) tumor molecular profiling with no pathologic variants in KRAS or NRAS or BRAF V600 mutations. If additional molecular profiling is completed (tissue or blood based testing) after receiving treatment for colon cancer and variants in KRAS or NRAS are found, those patients will be considered eligible for this study. Patients with BRAF V600 mutations are not eligible.
* Participants must not have known additional malignancy that is requiring systemic treatment. Participants taking hormonal treatments for breast or prostate cancer are still eligible.
* No major surgery within prior 2 weeks of treatment initiation (4 weeks if will be receiving bevacizumab).
* Urine protein less than 100 mg/dL if planning to receive bevacizumab.
* Blood pressure <160/90 if planning to receive bevacizumab.
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to panitumumab or cetuximab, including known severe hypersensitivity reactions to monoclonal antibodies. No history of allergic reactions to 5-Fluorouracil, irinotecan, leucovorin or bevacizumab if the participant will be receiving that agent in this study.
* Participants must have no metastatic cancer lesions greater than 3.5cm in diameter. Any number of metastatic lesions will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) at 6 months for Cohorts A and B | 6 months
  The disease control rate is the proportion of all subjects with stable disease (SD) for 8 weeks, or partial response (PR), or complete response (CR) according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).
Cohort C Progression Free Survival (PFS) | up to 4 years
  PFS will be defined as the duration (in months) from the date of study enrollment to date of disease progression (or death). If no progression (or death) event is observed during the follow-up period of the study, then PFS will be censored at the last date of follow-up per standard RECIST vs. 1.1 evaluation.

SECONDARY OUTCOMES:
Cohort A and B Progression Free Survival (PFS) | up to 4 years
  PFS will be defined as the duration (in months) from the date of study enrollment to date of disease progression (or death). If no progression (or death) event is observed during the follow-up period of the study, then PFS will be censored at the last date of follow-up per standard RECIST vs. 1.1 evaluation.
Cohort A, B, and C Objective Response Rate (ORR) | up to 1 year
  Objective responses which will include all confirmed complete responses (CR) and confirmed partial responses (PR) determined as per RECIST v1.1 on treatment with panitumumab in metastatic, left-sided, non-bulky colorectal cancer.
Type and Severity of Toxicities | up to 1 year (adverse events collected to 30 days post treatment)
  Toxicities will be graded using the most recent version of the CTCAE criteria. Toxicities will be summarized by type and severity in tabulator format.
Rate of Retreatment with EGFRi for Cohorts A and B | up to 4 years
  The rate of retreatment with EGFRi will be defined as the proportions of all eligible subjects who are retreated with EGFRi among all eligible subjects.
Cohort A, B, and C Overall Survival (OS) | up to 4 years
  OS will be defined as the duration (in months) from the date of study enrollment to the date of death (of any case). If no death event is observed during the follow-up period in a subject, then OS for that subject will be censored at the date of the last known survival status.

OTHER OUTCOMES:
Change in Participant Derived Organotypic Spheroid Response over baseline | baseline, post treatment (up to 1 year)
  To determine the ability of patient-derived colorectal cancer organoids to predict clinical response to EGFR inhibition, participant derived organotypic spheroids will be grown from biopsy at baseline assessment and compared to clinical response from EGFR inhibitor. This measure will a percentage change from the baseline.
Circulating Tumor DNA (ctDNA) at time of Progression | 1 month (cycle 1, day 1 of 28 cycle), 4 months (cycle 3, day 1 of 28 day cycle), up to 1 year (30 days post treatment)
  To evaluate ctDNA for early markers predictive of clinical resistance, ctDNA will be evaluated for subclonal alterations at the time of clinical disease progression and compared to repeat tissue biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Deming, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No